CLINICAL TRIAL: NCT07366242
Title: Prognostic Value of Dihydroorotate Dehydrogenase (DHODH) Expression in High-Grade Serous Ovarian Carcinoma: A Comparative Study Between Neoadjuvant and Adjuvant Chemotherapy Settings
Brief Title: Prognostic Value of (DHODH) Expression in (HGSOC): A Comparative Study Between Neoadjuvant and Adjuvant Chemotherapy Settings
Acronym: HGSOC
Status: Not yet recruiting | Type: Observational
Sponsor: Heba Ahmed Mohamed (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Heba Ahmed Mohamed, demonstrator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: DHODH in HGSOC; assiut university (Other: assiut university)
Record Dates: First submitted 2026-01-10; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HGSOC
MeSH Terms: interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A chemo naive and Group B neoadjuvant group: Group A (Chemo-naïve group) 36 Patients who underwent primary debulking surgery (PDS) followed by adjuvant platinum-based chemotherapy.
  Group B (Neoadjuvant group) 36 Patients who received 3-4 cycles of platinum-based neoadjuvant chemotherapy followed by interval debulking surgery (IDS).
  Interventions: Other: Immunohistochemical (IHC) assessment of DHODH expression; Other: No interventions as it is observational study
- Group A (Chemo-naïve group) 36 Patients and Group B (neoadjuvant) group: Group A (Chemo-naïve group) 36 Patients who underwent primary debulking surgery (PDS) followed by adjuvant platinum-based chemotherapy.
  Group B (Neoadjuvant group) 36 Patients who received 3-4 cycles of platinum-based neoadjuvant chemotherapy followed by interval debulking surgery (IDS).
  Interventions: Other: Immunohistochemical (IHC) assessment of DHODH expression; Other: No interventions as it is observational study

INTERVENTIONS:
Other: Immunohistochemical (IHC) assessment of DHODH expression — Comparative analysis of DHODH expression in adjuvant and neoadjuvant groups and correlate its expression with clinical outcomes
Other: No interventions as it is observational study — No interventions as itis observational study

SUMMARY:
* To compare DHODH protein expression in HGSC tissues from patients undergoing Primary Debulking Surgery (PDS - Chemo-naive) versus Interval Debulking Surgery (IDS - Post-NACT).
* To evaluate the association between DHODH expression and the degree of chemotherapy response (using the Chemotherapy Response Score - CRS for NACT cases).
* To determine the prognostic value of DHODH expression in predicting Platinum-Free Interval (PFI) ,Progression -Free Survival (PFS) and Overall Survival (OS) across both groups.

DETAILED DESCRIPTION:
High-grade serous ovarian carcinoma (HGSC) is the most aggressive and lethal subtype of epithelial ovarian cancer, accounting for nearly 70% of ovarian cancer-related deaths worldwide (1). Despite initial sensitivity to platinum-based chemotherapy, the majority of patients eventually develop chemoresistant disease, leading to recurrence and poor long-term survival (2). The biological mechanisms underlying platinum resistance remain incompletely understood, but increasing evidence indicates that metabolic reprogramming and redox adaptation play a central role in tumor cell survival under therapeutic stress (3).

Ferroptosis is a regulated form of cell death driven by iron-dependent lipid peroxidation, and it has recently emerged as an important vulnerability in cancer cells exposed to chemotherapy (4). Cancer cells that survive platinum-based therapy frequently upregulate antioxidant and lipid-repair systems that protect them from ferroptotic death (5). Among these systems, dihydroorotate dehydrogenase (DHODH), a mitochondrial enzyme involved in de novo pyrimidine biosynthesis, has been identified as a key suppressor of mitochondrial lipid peroxidation and ferroptosis (6).

DHODH is localized on the inner mitochondrial membrane and catalyzes the oxidation of dihydroorotate to orotate, coupling pyrimidine synthesis to the mitochondrial respiratory chain (7). Recent work has shown that DHODH acts in parallel with glutathione peroxidase-4 (GPX4) to protect cells from ferroptosis, particularly within the mitochondrial compartment (8). Inhibition of DHODH sensitizes cancer cells to oxidative damage and restores ferroptotic cell death, especially in tumors with high mitochondrial metabolism.

In ovarian cancer, platinum resistance has been linked to enhanced mitochondrial function, redox buffering, and metabolic plasticity ( 9). Neoadjuvant chemotherapy (NACT), which is increasingly used in advanced HGSC, exposes tumor cells to intense oxidative and genotoxic stress prior to surgical removal (10). This creates a strong evolutionary pressure favoring tumor clones capable of surviving chemotherapy-induced metabolic and redox stress.

However, the expression and clinical significance of DHODH in HGSC, particularly in the context of neoadjuvant chemotherapy exposure, has not been systematically investigated. No studies have directly compared DHODH expression in chemo-naïve primary debulking surgery (PDS) specimens versus post-NACT interval debulking surgery (IDS) specimens, nor correlated DHODH with chemotherapy response and survival outcomes. Understanding whether NACT selects for DHODH-high, ferroptosis-resistant tumor cells could provide novel insights into platinum resistance and identify a new therapeutic vulnerability in HGSC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade serous ovarian carcinoma
* Availability of adequate FFPE tumor tissue
* Known treatment modality (PDS or IDS)
* Available clinical follow-up including platinum-free interval and survival data

Exclusion Criteria:

* Non-serous histological subtypes
* Low-grade serous carcinoma
* Inadequate tissue for immunohistochemistry
* Missing clinical or follow-up data

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Archived formalin-fixed paraffin-embedded (FFPE) tissue blocks from patients diagnosed with high-grade serous ovarian carcinoma will be retrieved from the pathology archives
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
DHODH expression and patient survival | from diagnosis up to last follow up or death ( up to 96 months).
  To evaluate the prognostic impact of DHODH expression in high-grade serous ovarian carcinoma by assessing its correlation with survival outcomes (overall survival and/or progression-free survival) and comparing patients treated with neoadjuvant versus adjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No